CLINICAL TRIAL: NCT07017608
Title: Inspiratory Work of Breathing Before and After Extubation
Acronym: INTEGRATION
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Ewan Goligher, Ewan C Goligher, MD, PhD, University Health Network, Toronto
Other Study IDs: 19-5879
Record Dates: First submitted 2025-05-23; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Lung Transplant; Complications; Ventilator-Induced Lung Injury; Ventilator Associated Pneumonia
MeSH Terms: conditions — Ventilator-Induced Lung Injury; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Critically ill patients who (1) are not able to maintain their airway, (2) cannot breathe on their own, or (3) both, are ones who often require tracheal intubation and support from a breathing machine (mechanical ventilator). When the patient is ready to be liberated from the mechanical ventilator because the initial insult for intubation has been resolved, the patient is screened using the readiness to wean test in preparation for extubation. As the patient passes this screening, a spontaneous breathing test (SBT) is initiated. Currently, there are many debates surrounding which SBT technique is most favorable. At Toronto General Hospital, the clinical team uses a zero-end expiratory pressure (ZEEP) trial. Once the patient successfully passes their SBT they are then extubated.

The patient will undergo a spontaneous breathing trial of continuous positive airway pressure (CPAP) of 5 cmH2O and ZEEP, in which time the investigators will be using a new technology called electrical impedance tomography (EIT), to study and compare the end expiratory lung volume (EELV); investigators will use an esophageal catheter to measure and monitor pressures in the lung, and also assess the patient's work of breathing. This will be repeated once the patient has been extubated safely.

DETAILED DESCRIPTION:
Detailed Description:

Many patients in intensive critical care require mechanical ventilation. Once the underlying reasons for intubating critically ill patients have been addressed, healthcare providers aim to allow patients to return to breathing spontaneously and to safely remove the endotracheal tube (ETT) at the earliest appropriate time. Unnecessarily delaying the removal of the ETT (extubation) may cause diaphragm muscle weakening or introduce ventilator induced pneumonia (VAP), ventilator induced lung injury (VILI) and ventilator induced diaphragm dysfunction. Thus, it is important to determine when a patient is ready to be weaned from mechanical ventilation in a timely manner.

Spontaneous breathing trials (SBTs) can be used to aid in assessing a patient's readiness for extubation. There is currently no clear consensus on which technique is the most beneficial as there are uncertainties about how different SBT strategies impact both gas exchange and the work of breathing (WOB) before and after extubation. At Toronto General Hospital (TGH), patients are placed on a zero positive end expiratory pressure (ZEEP) SBT trial. It has been argued that the resistance from ETT increases WOB while a patient is on ZEEP, and this added effort may be eased through the use of low levels of pressure support or CPAP, which could potentially improve the success of extubation processes. Additionally, maintaining some amount of positive end expiratory pressure (PEEP) during SBT might improve oxygenation and WOB.

This study aims to understand how the zero positive end expiratory pressure (ZEEP) trial affects lung function and breathing effort in lung transplant patients who require mechanical ventilation in the ICU. The use of tools such as Esophageal and gastric balloon (NutriVent, Sidam, Mirandola, Italy), EIT (Drager PulmoVista 500), Pneumotachograph, FluxMed respiratory monitor, and Respiratory muscle ultrasound will be used to measure lung function, respiratory mechanics, muscle function, arterial blood gas, gastric pressure and esophageal pressure.

After enrolling 27 participants, this study has been amended to address an additional new objective - the validation of non-invasive occlusion maneuvers to estimate expiratory muscle pressure. Expiratory activity is a phenomenon that can provide important insights during mechanical ventilation and during an SBT trial. EELV might decrease due to expiratory muscle activity, possibly impairing gas exchange and increasing lung elastance due to collapse. Currently, the use of a gastric balloon is the gold standard method to assess expiratory effort and enable quantification of expiratory muscle pressure by expiratory variation of gastric pressure (∆Pga). However, the gastric balloon is an invasive tool that presents several downsides, as a high cost and the need for expertise in balloon calibration and waveform analysis. This highlights the need for non-invasive methods to detect and quantify expiratory muscle activity. The ability of occlusion maneuvers to detect presence of expiratory muscle effort measured with the gold standard (gastric pressure) will be assessed with receiver operating characteristic curves. A total of 40 patients will be enrolled to address this objective, in addition to the 27 patients already enrolled, for a total of 67 patients. Of the first 27 patients enrolled, only 15 underwent study procedures. Going forward, a patient will be considered enrolled if they undergo study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients intubated and ventilated

Exclusion Criteria:

* Contraindication for esophageal catheter insertion: upper gastrointestinal surgery within prior 6 weeks, actively bleeding esophageal varices
* Bronchopleural fistula
* Contraindication for electrical impedance tomography: chest burns, skin lesions in the thorax, chest wall bandaging limiting electrode placement, unstable spinal lesions or fractures
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients admitted to the medical surgical intensive care unit (MSICU) at Toronto General Hospital (TGH) requiring invasive mechanical ventilation, after obtaining consent. Inclusion will be stratified in a 1:1 ratio between lung transplant and non-transplant patients.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in end-expiratory lung volume (EELV) between the varying conditions (CPAP 5, ZEEP, and post-extubation). | Up to 30 minutes after extubation
  End-expiratory lung volume is assessed using Electrical Impedance Tomography (EIT) and expressed in milliliters (mL) across all three conditions:
  1. CPAP 5 cm H₂O
  2. ZEEP (Zero End-Expiratory Pressure)
  3. Post-extubation
Discriminative ability of occlusion maneuvers to detect expiratory muscle effort | Up to 30 minutes after spontaneous breathing trial initiation
  The ability of occlusion maneuvers to detect presence of expiratory muscle effort, measured with the gold standard (gastric pressure), will be assessed with receiver operating characteristic curves.

CONTACTS AND LOCATIONS:
Overall Officials: Ewan Goligher, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No